CLINICAL TRIAL: NCT02296788
Title: Effects of Aerobic Exercise on Gut Microbiota (EGM) - P & F Ancillary Study (E-Mechanic)
Brief Title: Effects of Aerobic Exercise on Gut Microbiota
Acronym: EGM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study wasn't stopped. It wasn't started. Funding.
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2014-062
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Gut Microbiota
Keywords: Gut Microbiota
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Exercise Control (No Intervention): Healthy Living Control Group
- Aerobic Exercise Group (Experimental): 8 kcal/kg of body weight/week (KKW) (~900 kcal/wk)
  Interventions: Behavioral: Aerobic Exercise
- Aerobic Exercise Group 2 (Experimental): 20 KKW (~2250 kcal/wk)
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — The exercise expenditure goals were calculated by multiplying the participants' body weight by the exercise dose (8 or 20 KKW) divided by the number of sessions (3-5 sessions/wk). The speed and grade were monitored and documented to keep participant heart rate at 65-85% of tested VO2 peak and entered into ACSM equations for energy expenditure.
  Arms: Aerobic Exercise Group; Aerobic Exercise Group 2

SUMMARY:
In the present study, we seek to elucidate the effects of aerobic exercise on fecal microbiota following the aforementioned no exercise control group and two doses of aerobic exercise training (the exercise training spans ~24 wks) in a cross-sectional sample.

DETAILED DESCRIPTION:
We will collect ancillary data for the ongoing Examination of Mechanisms of exercise-induced weight compensation (E-Mechanic; RCT; Martin CK and Church TS Co-PI's; R01 HL 102166) to investigate the independent aim and hypothesis of this pilot and feasibility (P & F) grant examining if there are differences in colonic microbial populations from a fecal sample following supervised and controlled aerobic exercise.

The proposed study seeks to better understand the role of colonic microbial populations as a mechanism of change in body weight during aerobic exercise. E-Mechanic is examining the effects of 2 tightly controlled and supervised doses of aerobic exercise, and a no-exercise control group, on energy balance and body weight over 24 wks in overweight and obese persons. The two aerobic exercise doses were: 1) 8 kcal/kg of body weight/week (KKW) (~900 kcal/wk) and 2) 20 KKW (~2250 kcal/wk) compared to a no exercise control group. The low dose of exercise (8 KKW) represents the American College of Sports Medicine (ACSM) recommendation for overall health and the higher dose (20 KKW) the recommendation for weight loss and weight loss maintenance.

Aim 1 To investigate if colonic bacterial populations differ between the exercise groups and the healthy living control group following aerobic exercise.

It is hypothesized that participants in the exercise group will have different bacterial populations than those in the healthy living control group.

ELIGIBILITY:
Inclusion Criteria:

Participants are overweight or obese (BMI 25 ≥ kg/m2 and ≤ 45 kg/m2), not actively exercising > 20 min on ≥ 3 days/wk, weight stable, non-diabetic, non-smoker, and not have any major medical disorders including such as HIV, CVD, mental illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota | 1 year